CLINICAL TRIAL: NCT03741998
Title: Nasopharyngeal Airway Facilitate Transnasal Humidified Rapid Insufflation Ventilatory Exchange
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RenJiH[2018]011
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Hypoxia; Hypercapnia
MeSH Terms: conditions — Hypoxia; Hypercapnia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- THRIVE (No Intervention): Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) during induction using jaw-thrust maneuver.
- THRIVE with nasopharyngeal airway (Active Comparator): Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) during induction with nasopharyngeal airway.
  Interventions: Device: Nasopharyngeal airway

INTERVENTIONS:
Device: Nasopharyngeal airway — THRIVE with a regular nasopharyngeal airway.
  Arms: THRIVE with nasopharyngeal airway

SUMMARY:
For performing transnasal humidified rapid insufflation ventilatory exchange (THRIVE), jaw-thrust maneuver have to maintain to make sure the airway open and the CO2 clearance during apnoea. The objective of present study is to prove that nasopharyngeal airway facilitate THRIVE and no need jaw-thrust maneuver and maintain the similar PO2 and PCO2 during apnoea.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Undergoing surgery with general anaesthesia.
* Adult, >18 years old.
* American Society of Anesthesiology classification I-II.

Exclusion Criteria:

* Coagulation disorders or a tendency of nose bleeding
* An episode/exacerbation of congestive heart failure (CHF) that requires a change in medication, diet or hospitalization from any cause in the last 6 months
* Severe aortic stenosis or mitral stenosis;
* Cardiac surgery involving thoracotomy (e.g., coronary artery bypass graft (CABG), valve replacement surgery) in the last 6 months;
* Acute myocardial infarction in the last 6 months;
* Acute arrhythmia (including both tachycardia and bradycardia) with hemodynamic instability;
* Diagnosed COPD or current other acute or chronic lung disease requiring supplemental chronic or intermittent oxygen therapy);
* Increased intracranial pressure;
* ASA >II;
* Mouth, nose, or throat infection;
* Fever, defined as core body temperature > 37.5°C;
* Pregnancy, breastfeeding or positive pregnancy test;
* Emergency procedure.
* Patient with known or suspected difficult airway

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-12-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
The partial pressure of carbon dioxide (pCO2) | From start to end of THRIVE(20 minutes)
The partial pressure of oxygen(PO2) | From start to end of THRIVE(20 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Diansan Su, Dr., Study Director — Renji Hospital, School of Medicine, Shanghai Jiaotong University, Shanghai, China
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen L, Yang L, Tian W, Zhang X, Zhao Y, Huang L, Tian J, Zhang J, Wu J, Yu W, Su D. Transnasal Humidified Rapid Insufflation Ventilatory Exchange With Nasopharyngeal Airway Facilitates Apneic Oxygenation: A Randomized Clinical Noninferiority Trial. Front Med (Lausanne). 2020 Nov 27;7:577891. doi: 10.3389/fmed.2020.577891. eCollection 2020. PMID 33330535